CLINICAL TRIAL: NCT01843816
Title: The Effect of Body Shape on Tragus-Wall Measurement
Status: Completed | Type: Observational
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihal Ozaras, Associate professor, Vakif Gureba Training and Research Hospital
Other Study IDs: tragus-wall
Record Dates: First submitted 2013-04-22; First posted 2013-05-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Obesity
Keywords: Tragus-to-wall distance; obesity; body shape; height; weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy subjects: 18-65 aged healthy subjects who have no disorder that may disturb posture or erect position (inflammatory diseases, kyphosis, scoliosis, joint deformities)

SUMMARY:
Tragus-to-wall distance (TWD) measurements is a method to evaluate spinal mobility in ankylosing spondylitis (AS) patients and it also takes place in Bath Ankylosing Spondylitis Metrology Index (BASMI). Being obese or slim may affect TWD. As well as the person's losing or taking weight may lead wrong evaluations, in comparative studies, according to the height or weight uneven distribution of groups may affect the results. The aim of this study is to investigate whether the body shape affect TWD or not.

DETAILED DESCRIPTION:
Healthy volunteers between 18-65 ages who have no disorder that may disturb posture or erect position (inflammatory diseases, kyphosis, scoliosis, joint deformities)will be included into the study. A wall corner will be used as the measurement platform; the evaluated person will be positioned as described in BASMI. A rigid ruler will be placed form anterior superior iliac spine (SIAS) to the lateral wall, parallel to the back wall; a projection point will be determined and its distance from back wall will be measured (SIAS-WD). In the same position, projection point of the middle of the humerus head and back wall distance (shoulder-WD) and TWD also will be measured. The relationships between these parameters will be statistically assessed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18-65 ages

Exclusion Criteria:

* subjects with disorders that may disturb posture or erect position
* inflammatory diseases,
* kyphosis,
* scoliosis,
* joint deformities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects between 18-65 ages who have no disorder that may disturb posture or erect position (inflammatory diseases, kyphosis, scoliosis, joint deformities)
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The assessment of the effects of having different weight and body shape on Tragus-Wall Measurement | 15 months
  Volunteers between 18-65 ages who have no disorder that may disturb posture or erect position (inflammatory diseases, kyphosis, scoliosis, joint deformities) will be included into the study.Their height, weight, hip circumference and tragus-to-wall distance will be measured. The relationship between these measurements will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Ozaras, Ass.Prof., Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)